CLINICAL TRIAL: NCT00628407
Title: Effect of Gentle Sternal Chest Wall Pressure on Intrathoracic Pressure During Mechanical Ventilation in Children.
Brief Title: Effects of Sternal Wall Pressure in Children
Acronym: SWP
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Laerdal Medical (Industry)
Responsible Party: Vinay Nadkarni, MD, Children's Hospital of Philadelphia
Other Study IDs: 2006-10-5023
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Respiration, Artificial
Keywords: leaning; CPR; sternal pressure; incomplete release; chest compressions; pediatric
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol is a prospective, pilot, observational study in the Pediatric Intensive Care Unit (PICU), Progressive Care Unit (PCU) and the Operating Room (OR) settings at the Children's Hospital of Philadelphia (CHOP). We propose to observe, measure and report the effect of incremental gentle sternal pressure increases on intrathoracic pressure, and other surrogates of hemodynamic function, in stable mechanically ventilated children. This study will provide preliminary data to inform the resuscitation research community and assist development of evidence-based pediatric resuscitation guidelines in the future.

DETAILED DESCRIPTION:
Context: Survival outcome following cardiac arrest in children is poor, and recent evidence suggests that the quality of Cardiopulmonary Resuscitation(CPR) is critically important. Venous blood return to the thorax to refill the heart is essential for good quality CPR and critical organ perfusion. Adult cardiac arrest studies suggest that incomplete chest wall decompression (i.e. "leaning" on the sternum of the chest) during CPR affects intrathoracic pressure and impedes venous return. The consequence of "leaning" on the chest during CPR is increased intrathoracic pressure, which creates a "back-pressure" preventing optimal return of blood to the heart. The critical importance of manipulating positive and negative intrathoracic pressures during Cardiopulmonary Resuscitation (CPR) has been recently demonstrated in both animal and human studies. Food and Drug Administration (FDA) approved defibrillators with a force and depth sensor can monitor the depth, rate and complete release of sternal pressure during CPR. These FDA approved defibrillators have been introduced and implemented in the Pediatric Intensive Care Unit (PICU) at the Children's Hospital of Philadelphia (CHOP). These defibrillators can provide feedback on the force and amount of "leaning", but there is no data on the minimal amount of sternal pressure (or "leaning pressure") that affects intrathoracic or intravascular pressures or venous return to the heart. In addition, there is no data on how much force on the sternal pressure sensor (e.g. leaning on the sensor) begins to affect intrathoracic pressure in children. We propose to observe, measure and report the effect of incremental gentle sternal pressure increases on intrathoracic pressure, and other surrogates of hemodynamic function, in stable but critically ill and mechanically ventilated children. This study will provide preliminary data to inform the resuscitation research community and assist development of evidence-based pediatric resuscitation guidelines in the future.

Objectives: 1) To characterize the effect of gentle, incremental increases in sternal chest pressure on intrathoracic pressure in mechanically ventilated children. 2) To characterize the effect of gentle, incremental increases in sternal pressure on regional perfusion pressures, when existing catheters (arterial, central venous, intracranial) are present.

Study Design/Setting/Participants: This protocol is a prospective, pilot, observational study in the Pediatric Intensive Care Unit (PICU), Progressive Care Unit (PCU) and the Operating Room (OR)settings at the Children's Hospital of Philadelphia. The participants are a convenience sample of stable mechanically ventilated children from 6 months to < 8 years of age. A total of 20 patients will be enrolled, including a minimum of 10 with vascular catheters.

Study Measures: The primary outcome variable is the change in intrathoracic pressure with incremental increase in gentle sternal pressure, measured by the peak airway pressure detected at the proximal end of the tracheal tube during end inspiration. Secondary outcomes include additional measures of intrathoracic pressure (end inspiratory pressure, mean pressure, area under the curve over 15 seconds, plateau pressure). For patients with indwelling central venous, arterial or intracranial pressure monitors, perfusion pressure changes will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to < 8 years.
* Weight greater than 4.8 kg.
* Hemodynamically stable (defined by the Pediatric Critical Care Team, Anesthesiologists and Surgeons)
* Volume Limited Ventilation Mode on Conventional Mechanical Ventilator
* Vascular catheters in place (for at least 10 subjects)
* Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

* Patients with contraindication to gentle, direct chest wall pressure (e.g. fresh sternotomy, recent chest wall surgery, chest tube in place)

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any patient in the Pediatric Intensive Care Unit (PICU), Progressive Care Unit (PCU) and Operating Room (OR) settings involving stable, mechanically ventilated children in the Children's Hospital of Philadelphia.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Nadkarni, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Sutton RM, Niles D, Nysaether J, Stavland M, Thomas M, Ferry S, Bishnoi R, Litman R, Allen J, Srinivasan V, Berg RA, Nadkarni VM. Effect of residual leaning force on intrathoracic pressure during mechanical ventilation in children. Resuscitation. 2010 Jul;81(7):857-60. doi: 10.1016/j.resuscitation.2010.03.015. Epub 2010 Apr 20. PMID 20409628

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were screened from January 1, 2007-June 2, 2008 using the protocol inclusion and exclusion criteria. Any patient in the PICU (7 South or 7 East), Progressive Care Unit (PCU) and Operating Room (OR) settings involving stable but critically ill, mechanically ventilated children from 6 months to < 8 years of age.
Groups:
- Sternal Wall Pressure: Subjects that received gentle incremental sternal wall pressure.
Period: Overall Study
Arm/Group | Sternal Wall Pressure
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sternal Wall Pressure
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 2.2 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Sternal Force Associated With Change in Intrathoracic Pressure.
Description: The mean sternal force (measured in kg as a surrogate for Newtons [1kg = 9.81 newtons]) associated with a ≥2cm H2O peak endotracheal pressure (ETP) change.
Time Frame: per case
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sternal Wall Pressure
Number analyzed (Participants) | 13
kg | 2.8 (0.9)

ADVERSE EVENTS:
Arm/Group | Sternal Wall Pressure
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No